CLINICAL TRIAL: NCT06057298
Title: Organoids From Colorectal Peritoneal Metastases to Improve Cytoreductive Surgery and Patient-tailored Hyperthermic Intraperitoneal Chemotherapy (HIPEC)
Brief Title: Patient-tailored Hyperthermic Intraperitoneal Chemotherapy (HIPEC) for Colorectal Peritoneal Metastases (OrganoHIPEC)
Acronym: OrganoHIPEC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT 0006/21; RF-2019-12370456 (Other Grant/Funding Number: Italian Health Minister Ricerca Finalizzata)
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-09

CONDITIONS: Peritoneal Metastases From Colorectal Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cytoreductive surgery and patient-tailored Hyperthermic Intraperitoneal Chemotherapy (HIPEC) (Experimental): * Preliminary laparoscopic exploration of the whole abdominal cavity is performed to stage the peritoneal disease, and obtain samples of peritoneal tumor to confirm the diagnosis of colorectal peritoneal metastases, and develop tridimensional cell cultures (organoids).
  * Preoperative systemic chemotherapy (s-CT) is performed at the discretion of treating medical oncologists, according to current guidelines.
  * Cytoreductive surgery and patient-tailored hyperthermic intraperitoneal chemotherapy (HIPEC) is scheduled within 6 weeks and at least 4 weeks after the completion of preoperative s-CT (at least 6 weeks after the last administration of bevacizumab). Cytoreductive surgery is aimed at removing all the macroscopic tumor by means od peritonectomy procedures and organ resections, as needed.
  Interventions: Procedure: Patient-tailored hyperthermic intraperitoneal chemotherapy (HIPEC)

INTERVENTIONS:
Procedure: Patient-tailored hyperthermic intraperitoneal chemotherapy (HIPEC) — Patient-tailored HIPEC is performed by the closed-abdomen technique with the following drugs selected according to the results of the sensitivity tests on the organoid-based preclinical model:
  * Oxaliplatin 360 mg/mq for 30 min.
  * Oxaliplatin 200 mg/mq for 120 min.
  * Mitomycin-C 35mg/mq for 60 min.
  * Mitomycin-C 3.3 mg/mq/l of perfusate + cisplatin 25 mg/mq/l of perfusate for 60 min. (perfusate volume l. 4-6)

SUMMARY:
The objective of this clinical trial is to demonstrate that cytoreductive surgery and patient-tailored hyperthermic intra-peritoneal chemotherapy (HIPEC) will increase efficacy in controlling peritoneal disease. Tridimensional cell cultures (organoids) derived from colorectal cancer peritoneal metastases are used to select the most active drugs in an in vitro HIPEC model on individual-patient level, based on the hypothesis that resistance to drug(s) routinely used for intraperitoneal delivery can explain peritoneal relapse after combined treatment, depending on the individual tumor biology;

DETAILED DESCRIPTION:
This single-arm, single-center, open-label trial enrolls patients with limited and surgically resectable peritoneal metastases from colorectal cancer, no distant metastases, and no contraindication to major surgery. After signature of informed consent, patients undergo a preliminary laparoscopy to confirm diagnosis of peritoneal metastases, stage the disease, and obtain representative samples of peritoneal metastases. The investigators will use patient-derived organoids to select tailored hyperthermic intra-peritoneal chemotherapy (HIPEC) regimens in an in vitro model HIPEC. A set of candidate drugs suitable for intraperitoneal administration are tested on tumor-derived organoids under the same conditions as in the clinical practice (same drug combinations, concentration, exposure time, temperature). Different concentrations are tested to generate reproducible dose-response curves. Patients receive 3-6 month preoperative systemic chemotherapy with targeted agents, according to current guidelines. Those not experiencing disease progression during preoperative systemic chemotherapy will have cytoreductive surgery and HIPEC with drugs selected on the organoid-based preclinical model. Patients will undergo postoperative follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of peritoneal metastases from intestinal-type or mucinous colo-rectal adenocarcinoma, by histological/cytological confirmation.
2. limited to moderate peritoneal involvement: peritoneal cancer index (PCI) ≤ 20;
3. peritoneal disease potentially amenable to complete surgical cytoreduction;
4. no evidence of hepatic, extra-regional nodal, or extra abdominal metastases
5. World Health Organization (WHO) performance status ≤2;
6. willingness to undergo preliminary laparoscopy, perioperative s-CT, and post-operative follow-up;
7. signature of informed consent.

Exclusion Criteria:

1. active sepsis;
2. impaired cardiac function (history of previous heart failure or 40% ejection fraction);
3. impaired renal function (serum creatinine >1.5 normal value or creatinine clearance < 60 ml/min);
4. impaired liver function (aspartate aminotransferase, alanine aminotransferase, bilirubin > 1.5 normal value);
5. impaired bone marrow function (leukocytes <4000/mm3, neutrophils <1500/mm3, platelets <80000/mm3);
6. impaired lung function (diagnosis of severe chronic obstructive pulmonary disease or 50% forced expiratory volume at one second or 40% diffusion capacity of lung for carbon monoxide adjusted for age);
7. dehydropyrimidine dehydrogenase deficiency;
8. pregnancy or lactation in progress;
9. haemorrhagic diathesis or coagulopathy;
10. any other condition or comorbidity that prevents safe administration of systemic chemotherapy (e.g. severe diarrhea, stomatitis or ulceration in the mouth or gastrointestinal tract);
11. psychiatric or neurological conditions that preclude the procedures of the protocol;
12. any contraindication to laparoscopy;
13. known hypersensitivity to any of the chemotherapy agents used for HIPEC in the present study and/or to any of their excipients;
14. history of previous malignancies treated in the last three years, excluding cutaneous spinocellular carcinoma and/or basocellular carcinoma;
15. previous cytoreductive surgery and HIPEC

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2025-06-14 (Estimated); Study Completion 2025-06-14 (Estimated)

PRIMARY OUTCOMES:
One-year peritoneal metastasis-free survival | 12 months
  Proportion of patients who remain free of peritoneal metastasis at a time interval of one year from the date of the combined procedure of cytoreductive surgery and patient-tailored hyperthermic intraperitoneal chemotherapy (HIPEC)

SECONDARY OUTCOMES:
Feasibility of patient-tailored hyperthermic intraperitoneal chemotherapy (HIPEC) | 48 months
  Feasibility will be determined as the number of patients who have cytoreductive surgery and patient-tailored hyperthermic intraperitoneal chemotherapy (HIPEC) among the total number of patients selected to be included in the study who sign the informed consent form
Overall survival | 60 months
  Overall survival will be measured from the date of cytoreductive surgery and patient-tailored hyperthermic intraperitoneal chemotherapy (HIPEC) to the date of death for any cause or, for patients still alive at the date of the last available follow-up
Disease-free survival | 60 months
  Disease-free survival will be measured from the date of cytoreductive surgery and patient-tailored hyperthermic intraperitoneal chemotherapy (HIPEC) to the date of peritoneal metastasis diagnosis, systemic metastases or death.
Safety of cytoreductive surgery and patient-tailored hyperthermic intraperitoneal chemotherapy (HIPEC) | 48 months
  Proportion of patients who will suffer from postoperative complications after cytoreductive surgery and patient-tailored hyperthermic intraperitoneal chemotherapy (HIPEC)

CONTACTS AND LOCATIONS:
Overall Officials: Dario Baratti, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano, Italy
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
I confirm that we have a plan to make individual participant data (IPD) available to other researchers through publicly available database
Supporting Information: Study Protocol, CSR
Time Frame: after the completion of the study, for additional 60 months
Access Criteria: upon reasonable request to the principal investigator

REFERENCES:
- [Background] Varinelli L, Guaglio M, Brich S, Zanutto S, Belfiore A, Zanardi F, Iannelli F, Oldani A, Costa E, Chighizola M, Lorenc E, Minardi SP, Fortuzzi S, Filugelli M, Garzone G, Pisati F, Vecchi M, Pruneri G, Kusamura S, Baratti D, Cattaneo L, Parazzoli D, Podesta A, Milione M, Deraco M, Pierotti MA, Gariboldi M. Decellularized extracellular matrix as scaffold for cancer organoid cultures of colorectal peritoneal metastases. J Mol Cell Biol. 2023 Apr 6;14(11):mjac064. doi: 10.1093/jmcb/mjac064. PMID 36460033
- [Background] Lorenc E, Varinelli L, Chighizola M, Brich S, Pisati F, Guaglio M, Baratti D, Deraco M, Gariboldi M, Podesta A. Correlation between biological and mechanical properties of extracellular matrix from colorectal peritoneal metastases in human tissues. Sci Rep. 2023 Jul 27;13(1):12175. doi: 10.1038/s41598-023-38763-w. PMID 37500685

DOCUMENTS (1):
  • Study Protocol (2020-12-28): https://cdn.clinicaltrials.gov/large-docs/98/NCT06057298/Prot_000.pdf